CLINICAL TRIAL: NCT07044219
Title: The Effect of Chlorhexidine (0.5%) With Combination of Hyaluronic Acid on Postoperative Wound Healing After Lower Third Molar Removal: a Placebo Controlled Triple Blind Randomized Clinical Trial
Brief Title: The Effect of Chlorhexidine + Hyaluronic Acid on Postoperative Wound Healing After Lower Third Molar Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Balazs Soos, Participating investigator, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7613-PTE 2019.
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Dry Socket; Postoperative Infections
Keywords: alveolitis; dry socket; dehiscence
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curasept DNA ADS periodontal gel (Experimental)
  Interventions: Procedure: Third molar surgery
- Placebo gel wound dressing (Placebo Comparator)
  Interventions: Procedure: Third molar surgery

INTERVENTIONS:
Procedure: Third molar surgery — During the operation, after local anaesthetics (LIDOCAIN-ADRENALIN 20 mg/0,01 mg/ml) the same mucoperiosteal (sulcular flap without vertical incision) is raised. Bone removal happens with physio-dispenser driven surgical handpiece (60ml/min irrigation; 8.000-16.000 rpm) and tungsten carbide round drills. Tooth section is made where indicated. After tooth removal wound is rinsed with 10-20ml physiologic salt, the wound is closed with 4.0 monofil non-resorbable suture material and then gel test or placebo is injected with syringe and applicator tip into the wound and on the surface of the wound. Patient bites a gauze for 20 minutes.

SUMMARY:
Our aim is to evaluate chlorhexidine-hyaluronic acid containing gel on postoperative wound healing regarding impacted lower third molar surgery.

DETAILED DESCRIPTION:
This is a triple-blind, placebo-controlled randomized clinical trial. Sixty patients will be randomly assigned to two treatment groups: Arm 1 receives Curasept DNA ADS periodontal gel during impacted third molar removal, while Arm 2 receives a placebo gel. Patient allocation uses an electronic randomization system with a 1:1 ratio. Baseline characteristics are recorded at the first clinical visit. The surgical procedure includes local anesthesia, mucoperiosteal flap elevation, bone removal with a surgical handpiece, and wound closure with non-resorbable sutures. Test gel or placebo is applied post-tooth removal, and patients are monitored postoperatively for pain, swelling, and wound healing, including follow-ups on the third, seventh and fourteenth days. Data analysis will use descriptive and statistical methods to evaluate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* patients having lower impacted third molar
* impaction pattern Pell-Gregory II/A, III/A, I/B, II/B, III/B that means partially impacted, partially erupted teeth, where primary wound closure is usually not possible;

Exclusion Criteria:

* systemic disease (diabetes, steroids, antiresorptive therapy);
* allergy on gel's compounds;
* pregnancy;
* active or subacute local infection at third molar tooth (pericoronitis);
* poor oral hygiene (based on the presence of active caries and/or plaque index of 2-3)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing | From enrollment to the end of treatment at 2 weeks
  Scoring wound healing according to Inflammatory Proliferative Remodelling (IPR) Wound Healing Scale: 0-16: the smaller number indicates the poorer outcome

SECONDARY OUTCOMES:
Mouth opening | From enrollment to the end of treatment at 2 weeks
Subjective pain level | From enrollment to the end of treatment at 2 weeks
  Visual Analogue Scale (VAS) 0-10: the higher number indicates the more intense pain.
Face swelling | From enrollment to the end of treatment at 2 weeks
Taken analgesics (questionaire) | From enrollment to the end of treatment at 2 weeks
  Reported amount of taken analgesics: 400 mg ibuprofen in each 6 hours in the first 48 hours, and after that as needed, but maximum 400 mg ibuprofen/6 hours +/- 500 mg paracetamol/6 hours.

OTHER OUTCOMES:
Probing pocket depth | From enrollment to the end of treatment at 2 weeks
  second molar

CONTACTS AND LOCATIONS:
Overall Officials: József Szalma, Prof, PhD, DSc, Study Director — UPMS Dept. Dentistry, Oral and Maxillofacial Surgery
Locations (1):
- Dept. of Oral and Maxillofacial Surgery, UP, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No